CLINICAL TRIAL: NCT01784809
Title: Multimedia HIV/STI Prevention for Drug-Involved Female Offenders
Brief Title: The Multimedia HIV/STI Prevention for Drug-Involved Female Offenders
Acronym: Project WORTH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Center for Court Innovation (Other); Bronx Community Solutions (Unknown); New York City Department of Probation (Unknown); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Nabila El-Bassel, PhD, Willma and Albert Musher Professor of Social Work, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAD5608; R01DA025878 (NIH)
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: HIV; Sexually Transmitted Infections
Keywords: HIV; STIs; Condom Use; Criminal Justice; Drug Use
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Multimedia HIV/STI prevention (Experimental): Multimedia WORTH is a 4-session group based gender specific HIV and drug abuse prevention intervention.
  Interventions: Behavioral: Multimedia WORTH
- Traditional HIV/STI prevention (Active Comparator): Traditional WORTH is a 4-session group-based HIV/STI and drug abuse prevention intervention that covers the same content as Multimedia WORTH without the use of interactive videos, computerized assessments, and other audiovisual tools.
  Interventions: Behavioral: Traditional WORTH
- Wellness Promotion (Placebo Comparator): Wellness Promotion is a 4-session group based intervention that aims to improve diet, physical fitness and well-being which is designed as an attentional control condition.
  Interventions: Behavioral: Wellness Promotion

INTERVENTIONS:
Behavioral: Multimedia WORTH — The Multimedia WORTH intervention features the same core elements as the original version, but these core elements are translated into interactive tools and culturally tailored video vignettes designed to enhance group learning and individualized feedback. Participants will interact with Multimedia WORTH at two levels: (1) group materials will be delivered via computer projection onto a screen and (2) participants will complete individual activities and create journal logs tracking their progress on personalized goals on their personal user accounts using laptop computers. The computer multimedia support tool includes text, imagery, animations, audio and video in a format that guide the facilitator's delivery of the intervention. ***To view pilot features of the Multimedia WORTH intervention in development, please visit the following web address:
  http://ccnmtl.columbia.edu/projects/worth/presentation
  Arms: Multimedia HIV/STI prevention
Behavioral: Traditional WORTH — The basic format of each WORTH session remains consistent following a sequence of 5 steps: (1) an opening (quote, song, poem) which will provide a brief culturally relevant point of inspiration to engage participants (2) Check-in to review material from the previous session, and to discuss any incidents where participants engaged in risk behaviors and to acknowledge positive ways in which women used new skills to avoid HIV risk; (3) a discussion to raise awareness of links between IPV, drug-related activities, and HIV risks; (4) a skills-building component relevant to the discussion; and (5) review and update participant needs, homework assigned for skills-building at home, and a closing ritual. The WORTH intervention consists of four 2-hour group sessions that are led by a female facilitator.
  Arms: Traditional HIV/STI prevention
Behavioral: Wellness Promotion
  Arms: Wellness Promotion

SUMMARY:
The proposed study addresses a significant public health threat of Human immunodeficiency virus (HIV) and sexually transmitted infections (STIs) among drug involved women on probation, parole or other community supervision. This randomized controlled trial aims to test the efficacy of a multimedia version of a 4-session, gender-specific, integrated drug use and HIV/STI prevention intervention (Multimedia Women On the Road To Health (WORTH)) in increasing condom use and decreasing the incidence of sexually transmitted infections (STIs) among 420 drug-involved, female offenders in a large community court setting in New York City, compared to a non-media version of the same intervention (Traditional WORTH) and to a 4-session Wellness Promotion condition.

DETAILED DESCRIPTION:
While it is clear that women inmates in jails and prisons bear a high burden of Human immunodeficiency virus/Acquired Immunodeficiency Syndrome (HIV/AIDS), the effective development of prevention interventions for this high-risk group require an understanding of HIV risk context, sexual behaviors and attitudes for women while they are still in the community and before they become heavily involved in the criminal justice system. HIV prevention interventions must focus on women at early points of entry into the criminal justice system, when they are still in the community and at higher risk of engaging in unsafe sex and drug behaviors. This study focuses on a population of drug-involved women who have been arrested and given a court sanction, but are still living in the community.

ELIGIBILITY:
Inclusion Criteria:

* She is 18 or older.
* She is currently supervised by a criminal justice entity, such as a community court or probation.
* She reports engaging in unprotected vaginal or anal sex with a male partner in the past 90 days
* She reports any illicit drug use or binge drinking in the past 6 months.

Exclusion Criteria:In addition, potential participants will be ineligible if any of the following criteria are met:

* Ability to speak and understand English is not sufficient to participate in assessments or intervention sessions.
* The woman's sexual activity is limited to a monogamous relationship lasting more than 12 months, and she has not engaged in any of the additional HIV risk behaviors in the past 90 days:

  * Having sex with more than one partner
  * Having sex with a partner known or suspected to be HIV positive or an injection drug user (IDU)
  * Sharing injection drug use needles or equipment
* The woman is actively trying to get pregnant/have a baby.
* Inability to complete informed consent process due to a psychiatric or cognitive impairment.
* The participant was born male.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2009-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The proportion of condom protected acts of vaginal and anal intercourse | Up to 12 months

SECONDARY OUTCOMES:
Cumulative incidence of biologically confirmed STIs (Chlamydia, Gonorrhea and Trichomoniasis) | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nabila El-Bassel, Ph.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University School of Social Work, New York, New York, United States

REFERENCES:
- [Derived] Slavin MN, West BS, Schreiber-Gregory D, Levin FR, Wingood G, Martino S, Tzilos Wernette G, Black C, El-Bassel N. Correlates of Unmet Need for Modern Contraception Among Reproductive-Aged Women Involved in New York City Criminal Legal Systems. Womens Health Rep (New Rochelle). 2024 Feb 16;5(1):132-142. doi: 10.1089/whr.2023.0177. eCollection 2024. PMID 38404679
- [Derived] Hochstatter KR, Slavin MN, Gilbert L, Goddard-Eckrich D, El-Bassel N. Availability of informal social support and the impact on health services utilization among women in community corrections who engage in substance use and risky sexual behavior: New York City, 2009-2012. Health Justice. 2022 Feb 16;10(1):6. doi: 10.1186/s40352-022-00170-0. PMID 35171362
- [Derived] El-Bassel N, Gilbert L, Goddard-Eckrich D, Chang M, Wu E, Hunt T, Epperson M, Shaw SA, Rowe J, Almonte M, Witte S. Efficacy of a group-based multimedia HIV prevention intervention for drug-involved women under community supervision: project WORTH. PLoS One. 2014 Nov 5;9(11):e111528. doi: 10.1371/journal.pone.0111528. eCollection 2014. PMID 25372149